CLINICAL TRIAL: NCT06757179
Title: Evaluation of the Therapeutic Effect of a Formulation Based on Mullein, Thyme, Propolis, and Long-Chain Polyphosphates in Children Diagnosed with Acute Rhinitis
Brief Title: The ELYAR (Elysium Against Rhinitis) Project
Acronym: ELYAR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Federico II University (Other)
Responsible Party: Principal Investigator, Roberto Berni Canani, MD, PhD, Md, PhD, Principal Investigator, Federico II University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 178/23
Record Dates: First submitted 2024-12-23; First posted 2025-01-03 (Actual); Last update posted 2025-01-03 (Actual); Status verified 2025-01

CONDITIONS: Rhinitis Viral

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Supplement (Experimental): Elysium Naso Gola Supplement is a dietary supplement designed to soothe the upper respiratory tract, providing a range of benefits thanks to the properties of its natural ingredients. Its anti-inflammatory, antibacterial, antifungal, antiviral, antioxidant, and prebiotic activities suggest a comprehensive product for supporting respiratory health.
  Mullein promotes the functionality of the respiratory mucous membranes. Thyme supports nasal and throat well-being, aids in the fluidity of bronchial secretions, and has antioxidant properties.
  Interventions: Dietary Supplement: Elysium Naso Gola
- Placebo (Placebo Comparator): Placebo
  Interventions: Other: Placebo

INTERVENTIONS:
Dietary Supplement: Elysium Naso Gola — Elysium Naso Gola Supplement is a dietary supplement designed to soothe the upper respiratory tract, providing a range of benefits thanks to the properties of its natural ingredients. Its anti-inflammatory, antibacterial, antifungal, antiviral, antioxidant, and prebiotic activities suggest a comprehensive product for supporting respiratory health.
  Mullein promotes the functionality of the respiratory mucous membranes. Thyme supports nasal and throat well-being, aids in the fluidity of bronchial secretions, and has antioxidant properties.
  Arms: Supplement
Other: Placebo — Placebo
  Arms: Placebo

SUMMARY:
Acute rhinitis is an inflammatory process that primarily affects the nasal mucosa, with a high incidence in the pediatric population and a morbidity rate of 6-8 episodes annually during the first two years of schooling (1). It is one of the most common conditions causing discomfort and debilitation in children, compromising their quality of life, negatively affecting social interactions, school performance, and sleep quality. In most cases, the origin is viral and the course is seasonal, with higher incidence in the autumn and winter seasons (1).

More than 100 viral strains are known to be responsible for this condition, among which Rhinoviruses are considered the most widespread and contagious (2). Symptoms, which typically begin 1-2 days after infection, include nasal congestion, nasal breathing obstruction, rhinorrhea, sneezing, coughing, headache, malaise, and sometimes mild fever, with complete remission generally occurring within 8-10 days (2).

The therapeutic approach is exclusively symptomatic, mainly aimed at reducing nasal obstruction. Literature indicates that nasal irrigation with saline solution is the most useful treatment for cleansing the nasal passages, thinning nasal secretions, and allowing for easier elimination; in the presence of fever, antipyretics may be useful (3).

Given these premises, the aim of this clinical study was to evaluate the therapeutic efficacy of an isotonic saline solution containing mullein, thyme, propolis, and long-chain polyphosphates, which are known for their natural properties to promote nasal secretion fluidity, reduce inflammation, and improve the functionality of the upper respiratory mucosa (4). In addition, more recent pre-clinical data suggested that this formulation exerts an antiviral action characterized by inhibition of virus replication (Rhinovirus and SARS-CoV-2) and an anti-inflammatory action through modulation of NF-Kb signaling in cultured human nasal respiratory epithelial cells. These effects are also associated with antibacterial action thanks to mullein and thyme.

ELIGIBILITY:
Inclusion Criteria:

* Caucasian subjects of both sexes,
* aged between 4 and 14 years;
* diagnosis of acute rhinitis based on the presence of ≥3 of the following symptoms that had onset within the last 24 hours: rhinorrhea, nasal congestion, nasal obstruction, sneezing, pharyngodynia, cough;
* in addition to ≥1 of the following signs/symptoms: headache;
* fever; malaise; burning eyes; myalgia;
* written informed consent obtained from the parents of the participants and from the participants themselves if older than 6 years.

Exclusion Criteria:

* non-Caucasian ethnicity; age <4 and >14 years; known hypersensitivity/allergy to any component of the dietary supplement;
* previous diagnosis of severe nasal septal deviation or any other condition that could cause nasal obstruction, such as nasal polyps;
* history of nasal or sinus surgery that could affect symptom scores; use of antibiotics, corticosteroids, or antihistamines within 2 weeks prior to the study; participation in other studies;
* conditions that made compliance with the protocol unlikely.

Ages: 4 Years to 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 60 (Actual)
Dates: Start 2023-12-01 (Actual); Primary Completion 2024-07-01 (Actual); Study Completion 2024-07-31 (Actual)

PRIMARY OUTCOMES:
severity of symptoms - score of Italian Nasal Obstruction Symptom Evaluation | after 5 days of treatment
  The primary endpoint was to assess the therapeutic efficacy of "Elysium Naso-gola" in reducing the severity of symptoms in children with acute rhinitis after 5 days of treatment with the Italian Nasal Obstruction Symptom Evaluation (I-NOSE questionnaire). A validated closed-question questionnaire with 5 items was administered to each enrolled subject to evaluate acute rhinitis symptoms. Each question was scored from 0 to 4 (0 = no problem; 4 = severe problem). The total score was multiplied by 5 to obtain the NOSE score, which classified the severity of nasal obstruction symptoms as follows: mild (5-25 points), moderate (30-50 points), severe (55-75 points), extreme (80-100 points).

SECONDARY OUTCOMES:
nasal obstruction - score of Visual Analog scale | after 5 days of treatment
  Secondary endpoints were the evaluation of the therapeutic efficacy of "Elysium Naso-gola" in reducing nasal obstruction in children with acute rhinitis after 5 days of treatment using the Visual Analog scale (VAS) . The VAS for nasal obstruction was graded from 0 to 10 mm, where 0 corresponded to "no obstruction" and 10 corresponded to "complete obstruction" (converted from 0 to 100% obstruction).
complete resolution of acute rhinitis symptoms | after 10 days
  the evaluation of the therapeutic efficacy of "Elysium Naso-gola" on the total complete resolution of acute rhinitis symptoms after 10 days.

CONTACTS AND LOCATIONS:
Locations (1):
- Roberto Berni Canani, Naples, Italy

IPD SHARING:
Plan to Share IPD: Undecided